CLINICAL TRIAL: NCT07055061
Title: An ISO Principle-Based Music Intervention for Reducing Stress, Anxiety, and Depression
Acronym: ISO4SAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, Yue DING, Associate Research Fellow, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THU0420251002; 62101324 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Stress; Anxiety; Depression in Adults
Keywords: music intervention; emotion regulation; ISO principle
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISO Group (Experimental): Participants in this group will receive a music intervention based on the ISO principle. The playlists are designed to gradually shift emotional states by starting with music that matches the participant's current mood and progressing toward tracks that reflect the desired emotional state, aiming to promote stress reduction and emotional regulation.
  Interventions: Behavioral: ISO Principle Music Intervention
- Compensation Group (Active Comparator): Participants in this group will receive a music intervention based on the compensation principle. The playlists directly contrast the participant's current emotional state by immediately introducing music that represents the target mood (e.g., relaxing music for a stressed state), with the aim of counteracting stress and promoting emotional change.
  Interventions: Behavioral: Compensation Principle Music Intervention

INTERVENTIONS:
Behavioral: ISO Principle Music Intervention — Participants will receive music playlists designed according to the ISO principle, which involves matching the participant's current emotional state and gradually transitioning to music reflecting a desired mood. The intervention aims to reduce stress and support emotional regulation by guiding affective resonance through music progression.
  Arms: ISO Group
Behavioral: Compensation Principle Music Intervention — Participants will receive music playlists based on the compensation principle, where the music contrasts the participant's current emotional state by directly presenting tracks aligned with the desired emotional outcome (e.g., calm music for stressed mood). This approach seeks to counteract stress and shift affective states through musical contrast.
  Arms: Compensation Group

SUMMARY:
This study aims to evaluate the effectiveness of a music-based intervention, guided by the ISO principle, in reducing stress, anxiety and depression induced by work, family or others among adults. The ISO principle suggests that emotional regulation can be supported by gradually modifying the emotional characteristics of music to help individuals transition to a desired emotional state.

Participants in this study will be randomly assigned to either a music intervention group or a control group. The intervention group will receive personalized music playlists designed to help reduce stress, anxiety and depression. The control group will not receive any music intervention during the same period.

Outcomes will be measured using self-report questionnaires assessing stress, emotional state, and well-being. The study is designed to contribute to the development of accessible, non-invasive stress management tools using music as a behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

* Has completed education at the associate degree level or higher
* Has at least one year of stable full-time work experience
* Maintains a regular and stable daily routine

Exclusion Criteria:

* Current or recent use of medication or history of surgical treatment
* History of psychiatric disorders
* Hearing impairments
* Female participants who are currently pregnant or breastfeeding

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Occupational Stress | Baseline, pre-intervention, Day1; Post-intervention, Day 6; 1 week post-intervention, Day 13; 1 month post-intervention, Day 36.
  Measured by the Occupational Stress Inventory Revised - Personal Strain Questionnaire (OSIR-PSQ). Participants complete the questionnaire at baseline and post-intervention to assess levels of personal strain related to work stress.
  The total scores range from 40 to 200, with higher scores indicating greater occupational stress.
Anxiety | Baseline, pre-intervention, Day1; Post-intervention, Day 6; 1 week post-intervention, Day 13; 1 month post-intervention, Day 36.
  Assessed using the Self-Rating Anxiety Scale (SAS). Measures general anxiety symptoms before and after the intervention. The total scores range from 20 to 80, with higher scores indicating greater anxiety severity.
Depression | Baseline, pre-intervention, Day1; Post-intervention, Day 6; 1 week post-intervention, Day 13; 1 month post-intervention, Day 36.
  Assessed using the Self-Rating Depression Scale (SDS). Evaluates depressive symptoms at baseline and post-intervention. The total scores range from 20 to 80, with higher scores indicating greater depression severity.

SECONDARY OUTCOMES:
State Anxiety | Before and immediately after each intervention session (twice per day of Day 2 to 6)
  Measured by the subscale State Anxiety Inventory (SAI) of The State-Trait Anxiety Inventory (STAI) to assess situational anxiety immediately before and after music intervention sessions. The total scores range from 20 to 80, with higher scores indicating greater anxiety severity.
Perceived Stress | Before and immediately after each intervention session (twice per day of Day 2 to 6)
  Visual Analogue Scale (VAS) used to assess subjective feelings of stress at multiple time points during the study. The score ranges from 1 to 100, with higher score indicating greater subjective stressful feelings.
Valence, Arousal, and Dominance | Before and immediately after each music piece (9 times per day of Day 2 to 6)
  Self-Assessment Manikin (SAM) used to measure emotional valence, arousal, and dominance immediately after each music listening session. The score of each dimension ranges from 1 to 9. Higher score of valence indicates more positive emotion. Higher score of arousal indicates greater emotional intensity. Higher score of dominance indicates stronger control of emotion.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Department of Psychology of Tsinghua University, Beijing, Beijing Municipality
  - Tsinghua University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time. A plan for data sharing will be developed prior to study completion.